CLINICAL TRIAL: NCT03257592
Title: PET Imaging of Glial Activation in Psychotic Disease States
Brief Title: Positron Emission Tomography (PET) Imaging of Glial Activation in Psychotic Disease States
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00037683
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with Schizophrenia Disorder (Experimental): Patients with Schizophrenia Disorder will be imaged with [11C] DPA-713
  Interventions: Drug: [11C]DPA-713
- Patients with Bipolar Disorder (Experimental): Patients with Bipolar Disorder will be imaged with [11C] DPA-713
  Interventions: Drug: [11C]DPA-713
- Control (Experimental): Normal volunteers will be imaged with [11C] DPA-713
  Interventions: Drug: [11C]DPA-713

INTERVENTIONS:
Drug: [11C]DPA-713 — [11C]DPA-713 PET imaging

SUMMARY:
Many neurological diseases, including AIDS dementia, Alzheimer's disease and schizophrenia, involve an inflammatory component thought to specifically involve glial cell activation. The Investigators has been concerned with the development of tools for noninvasive imaging of inflammatory processes in psychotic disease. Here, the investigators aim to use PET-based neuroimaging with carbon-11 N,N-diethyl-2-(4-methoxyphenyl)-5,7-dimethylpyrazolo[1,5-a]pyrimidine-3-acetamide, ([11C]DPA)-713 to quantify regional distribution of translocator protein (TSPO), a putative marker of inflammation, in the brains of patients with schizophrenia and bipolar disorder, type I. The investigators will focus on patients in the early stages of disease (within first five years of onset of schizophrenia diagnosis and within first five years of first manis, respectively) to minimize the confounds of age-, chronic illness-, and medication- effects on our results.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers 18-65 years of age
* Patients diagnosed with recent onset schizophrenia (within 5 years of onset), 18-65 years of age
* Patients diagnosed with recent onset bipolar disorder (within 5 years of onset of first mania), 18-65 years of age
* screening laboratory tests will be obtained for subjects within a 10 day period prior to the PET study and the results must be within normal limits for gender and age. These tests will be repeated with a 7-day window following the PET study
* EKG conducted within 10 day period prior to the PET study. The EKG will be repeated within 7 days following the study.
* Subject agrees to return to the Hospital for a follow-up EKG and laboratory testing of blood and urine.
* For females of childbearing potential, negative serum pregnancy test within a 10 day period prior to PET study.

Exclusion Criteria:

* history of recent nosocomial infection,
* history of chronic neurological disorder, such as multiple sclerosis or epilepsy, or structural,central nervous system (CNS) abnormality such as stroke or arteriovenous malformation,
* history of head injury with loss of consciousness > 1 hour,
* history of active substance abuse as defined by substance abuse including alcohol abuse over the 6 months prior to the study,
* dependence on benzodiazepine medication
* contraindications to MRI scanning to include pacemakers, metallic implants/prosthesis or prohibitive claustrophobia, etc.
* contraindications to PET scanning to include pregnancy, etc. For females of childbearing potential, negative serum pregnancy test less than 10 days prior to PET study
* ECG demonstrating the patient is not in a sinus rhythm or is having acute ischemia.
* any medical condition that in the opinion of the study investigators would constitute a safety risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of ([11C]DPA)-713 PET brain imaging in patients with recent onset schizophrenia and in patients with recent onset of mania | within five years of onset of schizophrenia or within five years of first manic episode
  To determine regional brain uptake of this radioligand in patients with recent onset schizophrenia and in patients with recent onset of mania

SECONDARY OUTCOMES:
PET Imaging of microglial activation | 5 years
  To evaluate changes in activation of microglia in patients with acute schizophrenia and bipolar disorder relative to controls

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pomper, MD,PhD, Principal Investigator — Professor
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States